

Icahn School of Medicine at Mount Sinai Mount Sinai Beth Israel Mount Sinai Brooklyn The Mount Sinai Hospital Mount Sinai Queens New York Eye and Ear Infirmary of Mount Sinai Mount Sinai St. Luke's Mount Sinai West Program for the Protection of Human Subjects Institutional Review Boards Mount Sinai Health System One Gustave L. Levy Place, Box 1081 New York, NY 10029-6574 T 212-824-8200 F 212-876-6789 irb@mssm.edu icahn.mssm.edu/pphs

## Amendment IRB-17-01796 Charles Ascher-Walsh

## **Table of Contents**

| 1. Modification | 1 |
|----------------------------------|----|
| 2. Summary - Title | 2 |
| 3. Summary - Setup | 3 |
| 4. Summary - Background | 5 |
| 5. Research Personnel | 6 |
| 6. Sites | 7 |
| 7. Subjects - Enrollment | 8 |
| 8. Subjects - Populations | 9 |
| 9. Subjects - Participation | 10 |
| 10. Procedures - Narrative | 11 |
| 11. Procedures - Genetic Testing | 12 |
| 12. Procedures - Details | 13 |
| 13. Procedures - Compensation | 14 |
| 14. Consent - Obtaining Consent | 15 |
| 15. Consent - Documents | 16 |
| 16. Data - Collection | 17 |
| 17. Data - HIPAA | 18 |
| 18. Data - Storage | 19 |
| 19. Data - Safety Monitoring | 21 |
| 20. Financial Administration | 22 |
| 21 Attachments | 23 |

## 1. Modification

#### **Summary of the Modification Request**

I would like to give the control group a B12 vitamin prior to surgery to act as a placebo.

## **Justification for the Modification**

After consideration of both groups and discussion with Attendings, we feel it would be less biased if the control group received a by mouth pill prior to surgery. I am proposing a vitamin as the pill given to the control group. The B12 vitamin I am proposing is over the counter and in some people changes the color of urine to orange, similar to pyridium. Hence it will increase the placebo affect on the patient's end.

This Modification Changes

the Consent Document or
Information that May Affect
Subjects' Willingness to Continue
to Participate in the Research

Description of Changes in the Consent Document or Information that May Affect Subjects' Willingness to Continue to Participate in the Research

In the areas where is it stated that the control group will receive nothing, it will be changed to them receiving a vitamin.

Subjects Will Be Re-Consented or Yes Provided with the New Information

#### Proposed Plan to Re-Consent Subjects or to Provide Them with the New Information

The patients already enrolled as controls did not receive vitamin B12, and have completed the intervention of the study. Therefore, re-consent is not necessary.

## 2. Summary - Title

#### **Protocol Title**

A randomized control trial assessing pyridium for post-sling urinary retention

Principal Investigator Charles Ascher-Walsh

When the application is complete, it will be sent to the PI for submission When the application is complete, it will be sent to the PI for submission

Primary Department Obstetrics/Gynecology

When the application is complete, it will be sent to the PI for submission

Application Initiated By Annacecilia Peacher-Seaney

### **Lay Summary**

Patients with stress urinary incontinence have the option of undergoing surgical intervention with a midurethral sling to improve if not cure their incontinence. One of the major complications of this procedure is urinary retention postoperatively. If a patient is not able to void on their own postoperatively they are required to go home from the hospital with a foley for bladder rest, and return to the clinic in 2-3 days to attempt a void trial once again. At our institution the rate of urinary retention after midurethral sling requiring discharge with an indwelling foley is 25% of patients who undergo this procedure.

Pyridium is a medication widely used and of low risk to the subject. It is a urinary numbing medication often used in patients with urinary tract infections. At the discretion of the physician, medication is given prior to midurethral sling and/or other urogynecologic procedures requiring cystoscopy to confirm bilateral ureteral jet efflux. The most common medication administered in the past was indigo carmine, now that this medication is off the market. Physicians have been using alternatives for visualization of ureteral jets on cystoscopy such a methylene blue, fluorescein, or pyridium. In this study patients undergoing midurethral slings will be randomized to one of two groups. The first group will receive pyridium preoperatively; the second will receive one 100mcg tablet of vitamin B12 as a placebo pill. The main goal of the study is to assess whether the group of patients who receive pyridium preoperatively have a lower rate of urinary retention postoperatively versus the control group. The secondary goal of the study is short term postoperative pain.

IF Number IF2052990

## 3. Summary - Setup

Funding Has Been Requested /

Obtained

**Application Type** 

Request to Rely on Mount Sinai IRB

Research Involves Prospective Study ONLY

**Consenting Participants** Yes **Requesting Waiver or Alteration** No

of Informed Consent for Any

**Procedures** 

Humanitarian Use Device (HUD)
Used Exclusively in the Course of

**Medical Practice** 

Use of an Investigational Device to Evaluate Its Safety or Effectiveness

Banking Specimens for Future

Research

No

Nο

No

No

Cancer Related Research that Requires Approval from the Protocol Review and Monitoring

Committee (PRMC).

Is this Cancer Related Research? Cancer Related Research is defined as research that has cancer endpoints or has a cancer population as part of or all of its targeted population. This includes protocols studying patients with cancer or those at risk for cancer.

Clinical Trial Yes

\* A prospective biomedical or behavioral research study of human subjects that is designed to answer specific questions about biomedical or behavioral interventions (drugs, treatments, devices, or new ways of using known drugs, treatments, or devices).

\* Used to determine whether new biomedical or behavioral interventions are safe, efficacious, and effective.

Drugs / Biologics

gics No

- \* Drugs / Biologics That Are Not a Part of Standard Practice
- \* Controlled Substances
- \* Drugs / Biologics Supplied by the Research Sponsor or Purchased with Study Funds

Ionizing Radiation for imaging or therapy, including X-Ray, Fluoroscopy, CT, Nuclear Medicine, PET andor Radiation Therapy:

\* Purely for standard of care:

No

\* In frequency or intensity that exceeds what is necessary for

No

cheederd of care.

standard of care:

Hazardous Materials No

- \* Viral Vectors
- \* Plasmids
- \* Bacterial Artificial Chromosomes
- \* Toxic Chemicals, Potentially Toxic Medications, Carcinogens \* Autologous Cell Lines

Request Use of Clinical Research No **Unit Resources** 

# 4. Summary - Background

### **Objectives**

To assess if there is a statistically significant difference in urinary retention after midurethral slings for stress urinary incontience in a group that receives preoperative pyridium versus a control.

#### **Background**

The prevalence of pelvic floor disorders in the United States is estimated to be 24%, with 16% of women experiencing urinary incontinence. Pelvic floor disorders affect a significant amount of women, and this increases with age.(3) Approximately 30% of women in the United States undergo corrective surgery, with a majority including incontinence surgery. The frequency of diagnosis of urinary tract infection after a sling procedure is 34% in the first three months, and 50% in the first year following a sling procedure.(1) Patients who are discharged with an indwelling foley after midurethral sling placement, undergo a risk of urinary tract infection that reaches 30%.(2)

- 1. Anger JT, Litwin MS, Wang Q, et al. Complications of sling surgery among female Medicare beneficiaries. Obstet Gynecol. 2007;109:707-714.
- 2. Dieter AA, Amundsen CL, Visco AG, et al. Treatment for urinary tract infection after midurethral sling: a retrospective study comparing patients who receive short-term postoperative catheterization and patients who pass a void trial on the day of surgery. Female Pelvic Med Reconstr Surg. 2012; 18(3): 175-178.
- 3. Nygaard I, Barber MD, Burgio KL, et al. Prevalence of symptomatic pelvic floor disorders in US women. Jama. 2008;300: 1311-1316.

#### **Primary and Secondary Study Endpoints**

Primary outcome: To evaluate if there is a statistical difference in urinary retention postoperatively after midurethral sling placement in patients who receive preoperative pyridium versus patients who receive routine perioperative care.

Secondary outcomes: Pain after surgery.

Pain Visual analog scale with documented log of pain postoperatively (starting at 2hrs-ending at 8hrs)(Half life of pyridium 8hr).

Protocol Was Already Approved
by the Icahn School of Medicine at
Mount Sinai (ISMMS) Institutional
Review Board (IRB) Under a
Different Principal Investigator

Protocol Was Previously Submitted No to an External(non-ISMMS) IRB

# 5. Research Personnel

| Name/Department | Role/Status | Contact | Access | Signature<br>Authority | Phone | Email |
|---|---|---|---|---|---|---|
| Charles Ascher-<br>Walsh / Obstetrics/<br>Gynecology | Principal<br>Investigator / | | Signature<br>Authority | | | |
| Annacecilia Peacher-<br>Seaney / | CI / | | Signature<br>Authority | | | |
| John Andrew Fantl / | CI / | | Edit<br>Access | | | |
| Woojin Chong-<br>Kaufman / | CI / | | Edit<br>Access | | | |
| Janine Doneza / | CI / | | Edit<br>Access | | | |

# 6. Sites

Site Name The Mount Sinai Hospital

**Other External Site Name** 

**Contact Details** 

Approved

**Approval Document** 

**Funded By Mount Sinai** 

Other IRB

IRB-17-01796 Amendment Charles Ascher-Walsh

# 7. Subjects - Enrollment

Site Name The Mount Sinai Hospital

**Subjects To Be Enrolled** 

98

Total Number of Subjects to be Enrolled Across All Listed Sites Above (Auto Populated)

98


## 8. Subjects - Populations

#### **Inclusion Criteria**

Any female patient undergoing a midurethral sling surgery, regardless of concomitant pelvic reconstructive or gynecological surgery.

#### **Exclusion Criteria**

Patients with complications from surgery requiring indwelling catheter, bladder/urethral perforation requiring indwelling catheter, acute bleeding requiring indwelling catheter for accurate urine output calculation, patients undergoing concomitant surgery other than gynecological, preoperative voiding dysfunction defined as postvoid residual >150cc, or spinal anesthesia. Women who are pregnant, including women of childbearing age who test positive on preoperative urine pregnancy test.

Enrollment Restrictions Based Yes
Upon Gender, Pregnancy,
Childbearing Potential, or Race

**Justify Restriction(s)** 

As part of the urogynecology specialty, I am only interested in analyzing female patients undergoing midurethral slings for stress urinary incontinence.

Age Range(s) 18 to 64 Years, 65 Years and Over

Targeted Population(s) Adults - Patients

#### Other Aspects that Could Increase Subjects Vulnerability

None to be noted, if a patient declines randomized medication prior to surgery they will receive the same perioperative care as all other patients.

#### Safeguards to protect Subjects rights and welfare

The patients' rights and welfare will be protected to the same standards as all patients undergoing surgery by our Urogynecology department at Mount Sinai Hospital.

## 9. Subjects - Participation

#### **Duration of an Individual Subjects Participation in the Study**

Approximately 1-2 days, starting with day of surgery and ending with Visual Analog Score 2-8 hours postoperatively

#### **Duration Anticipated to Enroll All Study Subjects**

Approximately 9 months according to 3-5 midurethral slings being performed at Mount Sinai Hospital per week. This is taking into consideration patient volume and subjects meeting inclusion/exclusion criteria.

Estimated Date for the Investigators Within two years to Complete This Study

#### **Procedures for Subjects to Request Withdrawal**

A patient can withdraw completely from the study by informing the principal investigator. They can call and ask to speak to Dr. Ascher-Walsh at FPA, or they can email Dr. Ascher-Walsh or Dr. Peacher-Seaney and let us know of their wish to withdraw.

#### **Procedures for Investigator to Withdraw Subjects**

It is not anticipated that patients will be withdrawn from the study by the research team. If a patient undergoes a complication in surgery necessitating an indwelling foley, or undergoes spinal anesthesia for their procedure, they will be removed from the study. When the voiding trial cannot be performed as it should, because of these constraints, it will be explained to the patient that they may have been in the treatment arm and received pyridium, however, due to the exclusion criteria of the study, their data cannot be used towards conclusions for the study.

Participants Will Be Recruited Yes

Recruitment Method(s) Clinical Practice

#### **How Participants Will Be Identified**

Any patients that are being consented for a midurethral sling procedure at FPA will be asked if they would like to participate in the study.

During a patient's preoperative visit, they will be screened to see if they meet inclusion/exclusion criteria. If they do, we will discuss how a cystoscopy is performed at the end of a case including a mid-urethral sling to inspect for bladder injury and uretheral patency. It will be discussed what medications can be given to aid in visualization of ureteral jets, and how pyridium is one medication that is often used for this. Then we will discuss that we want to test this medication to see if it decreases risks of urinary retention postoperatively. Then we will ask if they are interested in participating in the study.

Who Will Initially Approach
Potential Participants

Study Personnel

#### **How Research Will Be Introduced to Participants**

The research team approaching the patient asking if they are interested in the study will either be the surgeon, or fellow who will be participating in their surgery. If it is the fellow, they will be meeting the patient at the preoperative visit and discussing the study with them, in addition to being involved in the patient's surgical history and physical. It will be discussed that pyridium at times is used as standard of care during a urogynecologic procedure for visualization of ureteral patency during cystoscopy. In this study it will also be used to assess if it decreases the rate of urinary retention after midurethral sling procedure.

#### **How Participants Will Be Screened**

Patients who are having a midurethral sling procedure, who have not previously undergone an anti-incontinence procedure will be asked if they would like to participate.

Patients will be asked if they would like to participate in the study if they meet inclusion and exclusion criteria.

## 10. Procedures - Narrative

### **Description of the Study Design**

This is a prospective randomized controlled trial. It will have two arms with 48 patients in each arm, a total of 98 patients. Patients will be randomized with a block randomization schedule generated by computerized random numbers using a 1:1 allocation to pyridium and vitamin B12 placebo. The study is powered to see a difference in incidence of urinary retention after midurethral sling using 25% as the historic control for our institution. Statistical sample size was based on a decrease in incidence to 5% in the pyridium arm. This is with 80% power and alpha 0.05.

## **Description of Procedures Being Performed**

This study will use two study groups. One group will be given Pyridium 200mg po one hour prior to surgery. The second group will receive one 100mcg vitamin B12 tablet as a placebo pill. Patients will be randomized to either study group. After the patient's surgery, including a midurethral sling, they will have an active voiding trial performed as described by Pulvino et al. The patient's bladder will be backfilled with 300cc of sterile saline. If they cannot tolerate 300cc, they will be filled to maximum capacity. They will be allowed 20 minutes to void. The patient must void greater than two thirds the volume that was instilled in the bladder to consider it a passed voiding trial. The timing of the voiding trial will be at the discretion of the surgeon, accounting for factors such as complexity of concomitant surgery, the patient being alert, ambulating, with tolerable pain.

### Description of the Source Records that Will Be Used to Collect Data About Subjects

The electronic medical record Epic will be used to gather demographic information about patients.

## Description of Data that Will Be Collected Including Long-Term Follow-Up

Demographics will be gathered on patients, including: age, race, BMI, preoperative urodynamics and/ or simple cystometrics, obstetrical and gynecologic history, medical and surgical history.

Surgical procedures performed, if a patient passed or failed their active voiding trial.

Visual Analog Scale with documented log of pain postoperatively (starting at 2hrs-ending at 8hrs)(Half life of pyridium 8hr).

Research Requires HIV Testing No

# 11. Procedures - Genetic Testing

Genetic Testing Will Be Performed No
Guidance and Policies > Future Use Data Sharing and Genetic Research


# 12. Procedures - Details

Surveys or Interviews Yes

Type of Instruments Being Used Standardized

**Names of Standardized Instruments** 

Visial Analog Scale for pain

Audio / Photo / Video Recording No

**Deception** No

**Results of the Study Will Be Shared** No with Subjects or Others


# 13. Procedures - Compensation

**Compensation for Participation** No


## 14. Consent - Obtaining Consent

Consent Process Adult Consent

#### Where and When Consent Will Be Obtained

The consent will be obtained during the patient's preoperative visit or at an earlier visit if a specific surgical plan has been discussed prior to the preoperative visit at FPA.

#### **Waiting Period for Obtaining Consent**

A patient has the option of deciding about participation in the study and returning to clinic with the signed consent prior to their surgical date.

SOP HRP-090 Informed Consent Yes

**Process for Research Is Being** 

Used

PPHS Worksheets, Checklists and SOPs

Process to Document Consent in

Will Use Standard Template

Writing

Non-English Speaking Participants Yes

Will Be Enrolled

What Languages Other Than English Will Be Used

Spanish

What Process Will Be Used Long Form

The consent document must be translated into the language of the potential subject, and approved by the IRB, before you can go through the consent process with the non-English speaking person. If, after the project is approved, a short form consent process is needed, please see the PPHS policy and submit a modification.

# 15. Consent - Documents

**Consent Documents** 

Type Version 6.6.17
Name Version 6.6.17

Upload IDEATE Version 6.6.17 clean.doc

Consent Templates


## 16. Data - Collection

Health Related Information Will Be Yes

Viewed, Recorded, or Generated

### Description of Health Information That Will Be Viewed, Recorded, or Generated

Age, race, BMI, preoperative urodynamics and/ or simple cystometrics, obstetrical and gynecologic history, medical and surgical history.

Surgical procedures performed, if a patient passed or failed their active voiding trial.

Non-Health Related Information Will No

**Be Viewed or Recorded** 

HIV / AIDS Related Information Will No

Be Viewed or Recorded

Data That Will Be Viewed, Yes

Recorded, or Generated Contains ANY of the Following Directly

**Identifiable Information** 

Will Be Viewed Name, Medical Record Number, Telephone

number, Email Address

Will Be Recorded Name, Medical Record Number

**Data Collection Sheet** 

A Data Collection Sheet is required if you are either performing a retrospective review, or your study meets the category of exempt 4 research, or your study meets the category of expedited 5 research. Please upload it here.

Data Collection Source(s) Participant, Medical Chart (Paper or

Electronic)

## 17. Data - HIPAA

Obtaining HIPAA Authorization Yes

How PHI Will Be Protected from Improper Use or Disclosure

PHI will be saved on the password protected Mount Sinai desktop of the principal investigator.

PHI Will Be Destroyed at the Yes

**Earliest Opportunity Consistent** 

with the Research

When and How PHI Will Be Destroyed

When statistical analysis is completed for this study, the PHI will be permanently deleted from the hard drive of the prinicipal investigator's computer.

PHI Will Be Shared No

## PI must attest to the following.

\* I assure that the protected health information (PHI) will not be disclosed to any other person or entity not listed on this form except where required by law or for the authorized oversight of this research project. If at any time I want to reuse this PHI for other purposes or disclose it to other individuals or entities I will seek approval from the IRB.

## 18. Data - Storage

#### Location Where Data Will Be Stored

The data will be stored on the password protected Mount Sinai desktop of the principal investigator.

How will the data be stored? With a Code That Can Be Linked to the

Identity of the Participant

**Research Personnel Responsible** 

for:

Charles Ascher-Walsh

**Accessing Data** Yes **Receipt or Transmission of Data** Yes **Holding Code That Can Be Linked** Yes

to Identity of Participants

Annacecilia Peacher-Seaney

**Research Personnel Responsible** 

for:

**Accessing Data** 

Yes

**Receipt or Transmission of Data** Yes Holding Code That Can Be Linked

to Identity of Participants

No

**Research Personnel Responsible** 

for:

John Andrew Fantl

No **Accessing Data Receipt or Transmission of Data** No **Holding Code That Can Be Linked** Nο

to Identity of Participants

**Research Personnel Responsible** 

for:

for:

Woojin Chong-Kaufman

Accessing Data No Yes **Receipt or Transmission of Data Holding Code That Can Be Linked** Nο

to Identity of Participants

**Research Personnel Responsible** 

Janine Doneza

**Accessing Data** No **Receipt or Transmission of Data** Yes **Holding Code That Can Be Linked** No

to Identity of Participants

**Duration Data Will Be Stored** 

Until statistical analysis of the study is complete.

#### Steps That Will Be Taken to Secure the Data During Storage, Use, and Transmission

The data will be kept on the hard drive of the principal investigator's password protected Mount Sinai desktop.

#### Power Analysis/Data Analysis Plan (Including Any Statistical Procedures)

This is a two arm randomized controlled trial aimed to compare the rate of post-operative urinary retention between subjects given pyridium versus a control group. The primary outcome is the incidence of urinary retention measured prior to hospital discharge.

The rate of urinary retention is expected to be 25% in the control group. The proportion of subjects experiencing a primary outcome event will be compared between the groups using a two-sided T-tests of proportions. Assuming the proportion of patients experiencing post-op urinary retention is 25% in the control group a sample size of 48 in each group would give 80% power to detect a 20 percentage point reduction in urinary retention in the pyridium group. Patients will be randomized using a 1:1 allocation to pyridium and control. The secondary analyses is considered

exploratory and will be tested at the 0.05 significance level.VAS scores (ranging from 1-10) will be collected at 2- 6 hours post-operatively. Median score between the groups will be compared using a Wilcoxon test.


IRB-17-01796 Amendment Charles Ascher-Walsh

# 19. Data - Safety Monitoring

More Than the Minimum Data No Safety Monitoring Will Be Done

The following minimum requirements apply to all projects, including retrospective reviews of medical records, use of tissue samples, and many minimal risk studies, such as observational and survey research. Because these minimum requirements apply to all studies, a specific written DSMP will not usually be required for projects that do not pose greater than minimal risk to subjects. The MSSM PPHS may alter the required level of monitoring if appropriate.

For all projects, the principal investigator must have a plan to assure that data integrity will be maintained during its collection, storage and analysis. All research projects must adhere to MSSM recommendations on the storage of research data. Loss of data containing identifiable information is reportable to the IRB within 5 business days. Any problems concerning the consent process and any subject complaints should be monitored by the investigator. Reports of such problems must be made at least annually. The discretion of the protocol director will guide the need to report these problems immediately or more frequently.

The principal investigator is, typically, the monitoring entity for the minimum DSMP. When a principal investigator is not a faculty member, the supervising faculty member must be responsible for the data and safety monitoring aspect of the protocol.

Will the Research Include Data No Coordinating Center Activities?

## 20. Financial Administration

This information will help the Financial Administration of Clinical Trials Services (FACTS) office determine whether a Medicare Coverage Analysis (MCA) is needed for the research study. If you have any questions while completing this form, please contact the FACTS office at (212) 731-7067 or FACTS@mssm.edu.

Clinical Research Study Category Investigator Initiated

## Payment Options:

- \* Option 1: No protocol-required services will be billed to patients or third-party payers. Does Not Need MCA
- \* Option 2: Protocol-required services (i.e., routine care services) will be billed to patients or third-party payers. Must Have MCA
- \* Option 3: Study is initiated and federally funded by a Government Sponsored Cooperative Group who will only pay for services that are solely conducted for research purposes and other protocol-required services (i.e., routine care services) will be billed to patients or third-party payers. Billing Grid Only Required, NO MCA
- \* Option 4: Study involves only data collection and has no protocol-required clinical services. Does Not Need MCA
- \* Option 5: Study is not described in any of the above options. Please describe the study and specify whether External Sponsor (i.e., industry, government, or philanthropic source) and/or patient/third party payer will pay for protocol required services. MCA MAY Be Required

Payment Option

Option 1

No MCA is needed per option selected above.

## Payment Option 1:

- \* Option 1A: Department/collaborating departments will act as internal sponsor paying for all protocol-required services and no protocol-required services will be billed to patients or third party payers.
- \* Option 1B: Study involves protocol-required clinical services and an External Sponsor (i.e., industry, government, or philanthropic source) will pay for all protocol-required services.

**Payment Option 1** 

Option 1A

# 21. Attachments

| Туре | Name | Version | Status | Filename | Uploaded Date |
|---|---|---|---|---|---|
| Consent - Consent | Version 9.26 | 1 | New | IDEATE Version 9.26 | 09/28/2017 |
| Document | | | | clean.doc | |